CLINICAL TRIAL: NCT01502878
Title: Nut Allergy Study: Improving Diagnosis And Treatment Of Nut Allergy
Brief Title: Nut Allergy Study: Double-blind Challenge and Oral Desensitization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Mika Juhani Mäkelä, MD, PhD, Chief Physician, Helsinki University Central Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HUCHT101060080; IAS11 (Registry Identifier: HUCH, Skin and Allergy Hospital)
Record Dates: First submitted 2011-05-27; First posted 2012-01-02 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Nut Allergy
Keywords: Nut allergy; Double-blind placebo-controlled (DBPC) oral nut challenge; Nut oral immunotherapy (OIT); Nut oral desensitization
MeSH Terms: conditions — Nut Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Nut challenge (Active Comparator): Double-blind placebo controlled oral challenge 5-50-200-1000 mg peanut or hazelnut protein, or placebo administered with 30 min intervals and 2 hour-follow-up after the last dose.
  Interventions: Dietary Supplement: Nut challenge
- Nut challenge: Placebo (Placebo Comparator): See intervention
  Interventions: Dietary Supplement: Nut challenge: Placebo
- Nut oral desensitization (Experimental): Patients who have moderate to severe immediate allergic reaction at peanut challenge and who enter the oral desensitization program receive peanut protein daily, from 0,1 mg to 800 mg peanut protein, maintenance dose 800 mg.
  Interventions: Dietary Supplement: Nut oral desensitization

INTERVENTIONS:
Dietary Supplement: Nut challenge — Nut powder made from non-roasted nuts and roasted banana mixed with oats yoghurt or chocolate pudding
  Other Names: Super nuts banan chips; Yosa oat yoghurt; Arla cowpower chololate pudding
  Arms: Nut challenge
Dietary Supplement: Nut challenge: Placebo — Dried banana mixed with oat yoghurt or chocolate pudding
  Other Names: Super nuts banan chips; Yosa oat yoghurt; Arla cowpower chololate pudding
  Arms: Nut challenge: Placebo
Dietary Supplement: Nut oral desensitization — Roasted peanut powder mixed with milk- and soy-free margarine
  Other Names: Old Virginia Byrd Mill Fat-Light roasted peanut; Keiju-margarine
  Arms: Nut oral desensitization

SUMMARY:
Nut sensitization in skin prick tests is common in areas, including Finland, where birch pollen is abundant. However, sensitization to nuts in skin prick test does not predict the possibility of allergic symptoms when nuts are ingested. In this study the investigators launch and perform double-blind placebo-controlled nut challenges and oral desensitization/ protocol to those with serious symptoms in the challenge. The efficacy and safety of the new oral desensitization program is the primary outcome. The effect of oral desensitization on bronchial hyperreactivity, eosinophilic airway inflammation, and quality of life are secondary outcomes.

DETAILED DESCRIPTION:
The investigators aim to improve nut allergy diagnosis by launching a new double-blind placebo-controlled nut (peanut, hazel nut, cashew) challenge protocol. The investigators also launch a specific oral tolerance induction (SOTI) protocol to nuts in serious nut allergy. This study takes place in the Helsinki University Skin and Allergy Hospital between May 2011 and December 2015. Inclusion criteria: age 6 to 18 years and suspected nut allergy (unclear anaphylaxis possibly caused by nuts, skin prick test to nuts ≥ 10 mm or specific-IgE ≥ 20 kU/L and have never eaten nuts, or avoids nuts and does not dare try nuts at home). Patients having uncontrolled asthma or other lung disease, having cardiovascular disease or other systemic disease, using beta-blockers, and having poor compliance, are excluded. Methods:The investigators perform skin prick tests to peanut, tree nuts and seeds, take a blood sample before the double-blind placebo-controlled food challenges (DBPCFC), and measure total IgE and specific-IgE to birch, peanut, hazel nut, allergen components Ara h 1, 2, 3, and 8, and Cor a 1 and 8. Then the serum samples are kept frozen for further component and immunologic analyses. The investigators put iv before the challenge. In DBPCFC the patients receive 5 mg, 50 mg, 200mg, and 1000mg nut protein mixt with placebo, or placebo every 30 minutes. The severity of the allergic reaction is estimated using a modified severity scale. The probability of severe/moderate reaction at low (<0.7 kU/L) and at increased (>0.7 kU/L) Ara h 2 and 8 concentrations is the primary end-point in the DBPCFC. The investigators also correlate the concentrations of Ara h 2 with the severity score. Patients with moderate or severe reaction in the challenge will be offered desensitization therapy "SOTI" using(pea)nut flour mixed with milk-free margarine. The first dose of 0.1 mg nut protein is given at hospital part of the up-dosing is made at home every 2 weeks. The patient takes an antihistamine 1 hour before each daily dose. An epinephrine autoinjector and prednisolone tablets are also prescribed for emergency use. The desensitization protocol takes 28 weeks and is personalized when needed. Exercise is avoided 1 hour following each dose. Before and after the SOTI the investigators measure food related quality of life using standardized questionnaires, and perform metacholine challenge and measure exhaled nitric oxid. After the SOTI the investigators take blood samples and perform DBPCFC again.

ELIGIBILITY:
Inclusion Criteria:

* sensitization in skin prick test or in serum nut-specific IgE
* unknown anaphylaxis suspected caused by nuts
* never eaten nuts
* if challenge positive with serious symptoms, OIT

Exclusion Criteria:

* active asthma and low lung function,
* pregnancy, cardiovascular or other disease that might worsen during the challenge and OIT

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 102 (Actual)
Dates: Start 2011-05; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Efficacy of nut oral desensitization | 7 months
  Change from baseline in the amount of nut (mg) tolerated in a double-blind placebo-controlled oral challenge at 1 month after the 6-month oral desensitization therapy.

SECONDARY OUTCOMES:
Effect of the treatment on quality of life | 7 months
  Change from baseline in Quality of life questionnaire square before and after the oral desensitization therapy
Effect of the treatment on bronchial hyperreactivity and airway inflammation | 1 year
  Change from baseline in bronchial hyperreactivity in metacholine challenge and in eosinophilic airway inflammation measured by multiple channel exhaled nitric oxid
Safety of nut oral desensitization therapy | 7 months
  Number of participants with adverse events as a measure of safety and tolerability
Effect of the treatment on eosinophilic airway inflammation | 1 year
  Change from baseline in exhaled nitric oxid concentration

CONTACTS AND LOCATIONS:
Overall Officials: Mika J Mäkelä, MD, PhD, Principal Investigator — Helsinki UCH
Locations (2):
- Finland (2):
  - Helsinki University Central Hospital, Skin and Allergy Hospital, Helsinki, Finland
  - Helsinki University Central Hospital, Skin and Allergy Hospital, Helsinki, Helsinki

REFERENCES:
- [Derived] Uotila R, Kukkonen AK, Greco D, Pelkonen AS, Makela MJ. Peanut oral immunotherapy decreases IgE to Ara h 2 and Ara h 6 but does not enhance sensitization to cross-reactive allergens. J Allergy Clin Immunol. 2017 Apr;139(4):1393-1396.e6. doi: 10.1016/j.jaci.2016.09.054. Epub 2016 Dec 1. No abstract available. PMID 27916627